CLINICAL TRIAL: NCT05756530
Title: The Experience of Affective Touch in Obesity: the Role of Social Anhedonia and Lifespan Experiences
Brief Title: The Experience of Affective Touch in Anorexia Nervosa
Acronym: AffTouch_AN
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 21C127
Record Dates: First submitted 2023-02-22; First posted 2023-03-06 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Anorexia Nervosa
Keywords: affective touch; social anhedonia; lifespan bodily contacts; Interpersonal relationships
MeSH Terms: conditions — Anorexia Nervosa; Anhedonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Right-handed women diagnosed with restricting type or binge-eating/purging type AN, according to the Diagnostic and Statistical Manual of Mental Disorders (5th Edition)'s criteria (DSM, American Psychiatric Association, 2013), will be consecutively recruited during their rehabilitative treatment at the Istituto Auxologico Italiano, IRCCS, San Giuseppe Hospital (Italy). Concurrent neurological, neurodevelopmental (e.g., autism), motor, somatosensory and/or psychiatric disorders will be the exclusion criteria, as well as the evidence of any skin-related condition possibly affecting sensitivity on the participants' forearm (e.g., eczema, scars)
  Interventions: Other: Affective touch paradigm
- Controls: Age-matched, right-handed, healthy women (i.e., with no history of eating disorders) will be recruited outside the hospital through personal contacts of the researchers and word-of-mouth.
  Interventions: Other: Affective touch paradigm

INTERVENTIONS:
Other: Affective touch paradigm — Affective touch paradigm: experimental stimuli will include the touch of a soft cosmetic, a hand, which will be both expected to resemble affective pleasant stimulations, and a plastic stick with a rounded tip, as a control (non-affective) condition. Two speeds of stimulation will be adopted i) slow affective stimuli delivered at 3 cm/s and fast non-affective stimuli, delivered at non-optimal speed (18 cm/s). An imagery version of the task will be also administered: blindfolded participants will be asked to image the touches on their left forearm.
  After each (actual or imagined) tactile stimulus, individuals will rate the experience level of pleasantness.
  As part of the protocol, they will fill out two psychological questionnaires, assessing the level of social anhedonia and the amount and characteristics of the lifespan experiences of affective touch in close relationships.

SUMMARY:
The aim of the present research will be to verify if the pleasantness of affective touch is comparable between women with AN and healthy women while measuring the level of social anhedonia and the lifespan experience of affective touch.

ELIGIBILITY:
Inclusion criteria:

* Right-handed
* diagnosis of restricting type or binge-eating/purging type AN, according to the Diagnostic and Statistical Manual of Mental Disorders (5th Edition)'s criteria (DSM, American Psychiatric Association, 2013).

Exclusion Criteria:

* Concurrent neurological, neurodevelopmental (e.g., autism), motor, somatosensory and/or psychiatric disorders
* Evidence of any skin-related condition possibly affecting sensitivity on the participants' forearm (e.g., eczema, scars).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants with AN were consecutively recruited during their rehabilitative treatment at the Istituto Auxologico Italiano, IRCCS, San Giuseppe Hospital (Italy).
  -
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Rating of subjective pleasantness | Baseline
  Behavioural outcome associated with the experimental paradigm: participants will be asked to rate the pleasantness of the tactile stimuli after each stimulation with a score ranging from zero not pleasant at all) to 100 (extremely pleasant).

SECONDARY OUTCOMES:
Social Anhedonia Score | Baseline
  Social anhedonia will be evaluated with the Anticipatory and Consummatory Interpersonal Pleasure Scale (ACIPS, Gooding and Pflum, 2014); this is a 17-item self-report measure of individuals' tendency to look forward to interactions with others (anticipatory interpersonal pleasure - 7 items) and experienced pleasure in social interactions (consummatory interpersonal pleasure - 10 items). The ACIPS is scored on a Likert scale ranging from 1 (very false for me) to 6 (very true for me); higher scores indicate higher anticipatory and consummatory interpersonal pleasure.the assessment
Affective experience Score | Baseline
  The lifespan experience of affective touch in close relationships will be assessed with the Tactile Biography questionnaire (TBIO, Beltrán et al., 2020). This includes a 29-item self-report measure scored on a Likert scale ranging from 1 (e.g., not at all true for me) to 5 (e.g., extremely true) that evaluate four independent components: the frequency of and satisfaction for affective touch i) in childhood/adolescence and ii) adulthood, iii) comfort with and iv) fondness for interpersonal touch in close relationships. However, the experience of affective touch in adulthood was not included in the analyses since most of our participants did not have long experience in adult relationships since their age. Three additional items allow the recording of the feelings experienced in bodily affective interactions, the presence of negative/unpleasant experiences involving interpersonal touch and the preference for giving and/or receiving affective touch.affective touch in close relationships.

CONTACTS AND LOCATIONS:
Overall Officials: Federica Scarpina, PhD, Principal Investigator — IRCCS Istituto Auxologico Italiano
Locations (1):
- IRCCS Istituto Auxologico Italiano - Ospedale San Giuseppe, Piancavallo, VCO, Italy